CLINICAL TRIAL: NCT00274157
Title: Functional Improvement Through Revascularization of the Extremities for Peripheral Arterial Disease (FIRE-PAD). Effects of Catheter-Based Revascularization on Functional Capacity, Quality of Life, and the Cardiovascular Risk Profile of Patients With Intermittent Claudication
Brief Title: FIRE-PAD: Functional Improvement Through Revascularization of the Extremities for Peripheral Arterial Disease
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Dr Heather Gornik, Cleveland Clinic
Other Study IDs: FIRE-PAD
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral Vascular Disease; Intermittent Claudication; Catheter-based Arterial Revascularization; Peripheral angioplasty; Peripheral stenting; Functional capacity; Quality of life
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Behavior
Behavioral: diet control, smoking cessation, exercize

SUMMARY:
The specific aims of the project are as follows:

To determine whether catheter-based revascularization procedures improve functional capacity and quality of life among patients with intermittent claudication.

To investigate whether improvements in walking ability result in a less sedentary lifestyle and improvement of the cardiovascular risk profile.

DETAILED DESCRIPTION:
Patients with intermittent claudication have decreased functional abilities and impaired quality of life [QOL]. In addition, peripheral arterial disease is associated with an increased risk of a life threatening cardiovascular event. Due to advances in endovascular technologies, peripheral revascularization procedures are now offered to a growing number of patients with lifestyle limiting claudication, rather than solely for the treatment of critical limb ischemia. Indeed, according to data derived from the National Health Discharge Survey, there was a 979% increase in the number of catheter-based revascularization procedures performed during the period 1995-2000. Despite well defined patency outcomes, the functional and QOL benefits of catheter-based revascularization procedures are largely undefined. In addition to improving leg symptoms and QOL, increasing walking ability among patients with claudication may lead to a less sedentary lifestyle and improvement of the cardiovascular risk factor profile. However, this relationship has not yet been demonstrated. The proposed project is a longitudinal cohort study that will follow patients with intermittent claudication for one year after a catheter-based revascularization procedure to measure changes in functional capacity, QOL, and cardiovascular risk factors. Patients will be evaluated at baseline and at 3 and 12 months following the procedure. A total of 60 patients will be studied over a three-year period. Functional parameters to be assessed will include treadmill walking distances, the 6-minute walk test, walking velocity, and self-assessed walking ability as determined by the Walking Impairment Questionnaire. Activity level during daily life will be assessed using a vertical accelerometer device, which will be worn by patients for a 7-day period at each time point. Quality of life will be assessed by the Short Form-36 Questionnaire and the Geriatric Depression Scale. Cardiovascular risk factors to be measured will include anthropomorphic parameters, blood pressure, lipids, markers of inflammation, homocysteine, and insulin-sensitivity. It is intended that data generated from this study will provide initial data to plan a multi-centered randomized clinical trial of best medical therapy and exercise training versus catheter-based revascularization for the treatment of lifestyle limiting claudication.

ELIGIBILITY:
Inclusion Criteria:• Males and female between 40 and 85 years of age

* subjects referred to The Cleveland Clinic Foundation for a catheter-based revascularization procedure as treatment of intermittent claudication
* Leg symptoms consistent with intermittent claudication for a period of at least 3 months
* Ankle-brachial index (ABI) in the leg to be revascularized must be < 0.90 or demonstration of post exercise fall in ABI to < 0.9 for subjects with aortoiliac disease
* Subjects scheduled for both aortoiliac and/or femoropopliteal revascularization procedures will be eligible
* Subjects with bilateral leg symptoms may be enrolled, as long as bilateral revascularization procedures are planned

Exclusion Criteria:

* • Vascular anatomy inappropriate for a catheter-based procedure on the basis of non-invasive studies

  * Critical limb ischemia (rest pain, non-healing ulcer, gangrene)
  * Contraindication to contrast arteriography
  * Vascular surgery or prior catheter-based vascular intervention within the preceding 6 months
  * Patients with suspected or confirmed graft stenoses or occlusions
  * Myocardial infarction or hospitalization for unstable angina, coronary artery bypass grafting or percutaneous coronary intervention, within the preceding one month
  * Stroke or transient ischemic attack within the preceding one month
  * Pregnancy or planned pregnancy during the one year of participation in the trial.
  * Any active chronic inflammatory condition,including autoimmune disorder or active malignancy.Subjects unable to walk, amputees, and subjects with a contraindication to treadmill exercise.
  * Patients with dementia or other significant cognitive impairment
  * Patients who are non-English speaking, (due to the need for subjects to complete standardized questionnaires)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Gornik, M.D. M.H.S., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States